CLINICAL TRIAL: NCT03214354
Title: A Phase II Pilot Study of Nonmyeloablative Conditioning Hematopoietic Stem Cell Transplantation in Children with Sickle Cell Disease Who Have a Matched Related Major ABO-Incompatible Donor (Sickle-AID)
Brief Title: Nonmyeloablative Stem Cell Transplant in Children with Sickle Cell Disease and a Major ABO-Incompatible Matched Sibling Donor
Acronym: Sickle-AID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tony H. Truong, Pediatric Hematologist/Oncologist, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRU-17-001
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease; Stem Cell Transplant Complications; Red Blood Cell Disorder; Pure Red Cell Aplasia
Keywords: sickle cell disease; stem cell transplant; red blood cell engraftment; nonmyeloablative; pure red cell aplasia
MeSH Terms: conditions — Anemia, Sickle Cell; Red-Cell Aplasia, Pure | interventions — Alemtuzumab; Whole-Body Irradiation; Sirolimus

STUDY DESIGN:
Intervention Model Description: Phase II pilot, non-randomized, prospective study to evaluate the safety and efficacy of a nonmyeloablative conditioning allogeneic stem cell transplantation for patients with sickle cell disease who have a matched related major ABO-incompatible donor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-myeloablative conditioning (Experimental): Non-myeloablative conditioning
  Interventions: Drug: Alemtuzumab; Radiation: Total Body Irradiation; Drug: Sirolimus

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab, Day -7 to -3. Dose: 0.2mg/kg/dose SC once daily x 5 days
  Other Names: Campath
Radiation: Total Body Irradiation — TBI 300 cGy on Day -2
  Other Names: TBI
Drug: Sirolimus — Sirolimus is used for GVHD prophylaxis

SUMMARY:
The aim of this study to evaluate the safety and efficacy of a nonmyeloablative conditioning regimen for allogeneic hematopoietic stem cell transplantation (HSCT) in pediatric patients with sickle cell disease (SCD) who have a matched related major ABO-incompatible donor. The nonmyeloablative regimen will use alemtuzumab, total body irradiation (TBI) and sirolimus for immune suppression. This study will expand the access of HSCT for patients with SCD who are currently not eligible because of donor restrictions.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a debilitating chronic blood disorder with multi-system end-organ damage that leads to morbidity and early mortality. The only cure for SCD is hematopoietic stem cell transplantation (HSCT), which given the risks with unrelated HSCT, is only an option for a minority of patients who have a matched sibling donor.

In the field of HSCT, blood group ABO incompatibility between donor and recipient is not a contraindication and several studies do not show compromised outcomes. However, in the context of nonmyeloablative (NMA) conditioning and major ABO-incompatibility, when the recipient has existing antibodies to donor red blood cells, pure red cell aplasia (PRCA) may occur.

This phase II pilot study will enroll SCD patients with a matched related major ABO-incompatible donor to determine the safety and efficacy of NMA-HSCT. Biological studies will include a plan to study and monitor red cell engraftment in this population to facilitate early detection and interventional measures to prevent and treat PRCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 12 months and < 19 years of age at the time of study enrollment.
* Patients must have sickle cell disease as defined by hemoglobin electropheresis, as follows:

  * homozygous Hb S disease (HbSS),
  * sickle-Hb C disease (HbSC),
  * sickle beta-plus-thalassemia (HbS/β+), or
  * sickle beta-null-thalassemia (HbS/βo)
* Patients must meet standard eligibility criteria to undergo HSCT, including but not limited to one or more of the following:

  * history of repeated (more than 1) bony (vaso-occlusive) crisis
  * history of stroke
  * elevated transcranial Doppler velocity not eligible for hydroxyurea, as per TWiTCH trial (ie. severe vasculopathy)
  * history of acute chest crisis or splenic sequestration crisis
  * history of priapism in males
  * history of osteonecrosis
  * pulmonary hypertension as documented by tricuspid regurgitation jet velocity (TRV) > 2.5 m/s on echocardiogram
  * red cell allo-immunization (≥ 2 antibodies) during long term transfusion therapy
* Sickle complications should be present despite the use of hydroxyurea, but this is not an absolute requirement, if the treating team considers the patient to be at high risk for further crisis episodes.

Exclusion Criteria:

* Patients who are unable to comply with or follow the study protocol.
* Patients with known hypersensitivity to sirolimus, its derivatives or to any of its components.

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of pure red cell aplasia (PRCA) | 6 months from enrollment
  Clinical definition: reticulocytopenia < 10x109/L (< 1%) lasting more than 60 days after HSCT, or Pathological definition: the absence of erythroid precursors in the marrow in the setting of adequate myeloid, lymphoid and megakaryocytic precursors

SECONDARY OUTCOMES:
RBC chimerism measured by peripheral blood flow cytometry | 12 months
  Peripheral blood for RBC chimerism on flow sorted erythroid precursor cells
RBC chimerism measured by bone marrow BFU-erythroid forming colonies | 2 months
  Bone marrow will be performed between Day +45 and +60
Primary graft failure | 6 weeks
  Measured by donor chimerism from peripheral blood and bone marrow
Secondary graft failure | 24 months
  Measured by donor chimerism in peripheral blood and bone marrow
Disease recurrence | 24 months
  Measured by peripheral blood Hb S level
Incidence and severity of acute GVHD | 100 days
  Acute GVHD grade will be accessed using modified CIBMTR criteria
Incidence and severity of chronic GVHD | 24 months
  Chronic GVHD will be accessed using the NIH consensus criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No